CLINICAL TRIAL: NCT03776097
Title: Non-interventional Long-term Follow-up Observation After Surgical Treatment of Peri-implantitis in Multicenter Post Market Clinical Follow-up (PMCF) Study 13.530.231
Brief Title: Long-term Follow-up Observation After Surgical Treatment of Peri-implantitis in Multicenter Post Market Clinical Study
Status: Completed | Type: Observational
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 23530231
Record Dates: First submitted 2016-08-08; First posted 2018-12-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Defect Fill.: Observational study of the patients that were treated with biomaterials at the surgery in the previous study
  Interventions: Other: observational study
- No defect Fill.observational: Observational study of the patients that were not treated with biomaterials at the surgery of te previous study
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational study

SUMMARY:
The objective of this non-interventional long-term follow-up observation is to evaluate the long-term sustainability of two surgical treatments of peri-implantitis with and without Geistlich Bio-Oss® and Geistlich Bio-Gide® from a previous study

DETAILED DESCRIPTION:
The study is a non-interventional long-term follow-up observation without any study specific procedure outside normal clinical routine. Patients from a previous study are selected to participate in this study within a standard maintenance Programm. Primary and secondary oucomes refer to the previous study

ELIGIBILITY:
Inclusion Criteria:

* Implant survival at the treated site from the previous study
* Written informed consent

Exclusion Criteria:

* Implant failure at the treated site
* Severe trauma to implant site causing removal of the implant since the last visit of previous study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from a previous study
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-12; Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Defect fill | 2 years after the start of the study
  The primary outcome measure will be the change of "bone levels"(defect fill) over 2 years starting 1 year after surgical Intervention as assessed from intra-oral radiographs. In particular, the distances between the most apical implant to bone contact level and a characteristic reference point being the same for all sets of radiographs will be measured. The distance equal to three implant threads (known for the implant system) will be measured with a specific Software. The deeper bone level at baseline will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Rasi, PhD, Study Director — Geistlich Pharma; Stefan Renvert, Principal Investigator — Kristianstadt University
Locations (1):
- Kristianstad University, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: Undecided